CLINICAL TRIAL: NCT06335004
Title: Valutazione Delle Vie "Glinfatiche" Utilizzando la Risonanza Magnetica Nelle Malattie Della Sostanza Bianca
Brief Title: Evaluation of Brain Waste Clearance Pathways Using Magnetic Resonance Imaging in Pediatric Patients With White Matter Diseases
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Other Study IDs: 926
Record Dates: First submitted 2022-05-05; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Glymphatic System; White Matter Disease; Pediatric Disorder; Perivascular Disease
Keywords: Glymphatic system; white matter disease; perivascular space; diffusion tensor imaging; gadolinium; rare disease
MeSH Terms: conditions — Leukoencephalopathies; Rare Diseases | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with white matter disease/healthy subjects: Patients with white matter disease due to genetic or acquired causes. MRI with or without intravenous gadolinium will be performed
  Interventions: Diagnostic Test: Magnetic resonance imaging
- Patients with no white matter disease: Patients undergoing MRI with or without gadolinium for clinical diagnostic purposes, with no known white matter disease.
  Interventions: Diagnostic Test: Magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: Magnetic resonance imaging — Patients will undergo a magnetic resonance imaging for clinical purposes to which additional sequences. Post gadolinium research sequences will be acquired only if intravenous gadolinium needs to be administered for clinical purposes.

SUMMARY:
The dilation of perivascular spaces can be the result of various etiopathogenetic processes. White matter atrophy can cause enlargement of these perivascular spaces (PVS) but also obstruction of fluid drainage systems (interstitial fluid, ISF) and metabolites, as evidenced by some recent studies. Focal stagnation of liquids and deposition of toxic material induce tissue hypoxia and neuroglial dysfunction. Dilation of PVS can be associated with changes in white matter and microhemorrhages. We want to study these etiopathogenetic phenomena by implementing specific MRI methods.

DETAILED DESCRIPTION:
Primary objective: the quantification of indirect magnetic resonance markers of altered waste drainage systems using validated scales in patients with white matter disease. Secondary objective: the evaluation of white matter alterations in relation to the known anatomical glymphatic pathways by analyzing both structural and diffusion data.

ELIGIBILITY:
Inclusion Criteria:

* patients with and without white matter disease
* patients willing to participate in research with signed consent form
* no age limit (results will be age matched)

Exclusion Criteria:

* unwilling to participate in research

Ages: 9 Months to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with white matter disease on T2 and FLAIR sequences are included in this study. New MR sequences that can further identify subtle signal intensity changes within these white matter lesions will allow to further characterise them. Some patients will require intravenous gadolinium as part of their diagnostic MR work-up. Research MR sequences will also be acquired after gadolinium admininstration to further improve characterisation of the composition of white matter lesions.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Extent of white matter lesions | once at recruitment
  T1 values of lesions
Number of perivascular spaces | once at recruitment
  count of perivascular spaces and total volume in disease population
Volume of parasagittal dural space | once at recruitment
  volume of parasagittal dural space in disease population

CONTACTS AND LOCATIONS:
Locations (1):
- Scientific Institute IRCCS Eugenio Medea, Bosisio Parini, Lecco, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wardlaw JM, Smith EE, Biessels GJ, Cordonnier C, Fazekas F, Frayne R, Lindley RI, O'Brien JT, Barkhof F, Benavente OR, Black SE, Brayne C, Breteler M, Chabriat H, Decarli C, de Leeuw FE, Doubal F, Duering M, Fox NC, Greenberg S, Hachinski V, Kilimann I, Mok V, Oostenbrugge Rv, Pantoni L, Speck O, Stephan BC, Teipel S, Viswanathan A, Werring D, Chen C, Smith C, van Buchem M, Norrving B, Gorelick PB, Dichgans M; STandards for ReportIng Vascular changes on nEuroimaging (STRIVE v1). Neuroimaging standards for research into small vessel disease and its contribution to ageing and neurodegeneration. Lancet Neurol. 2013 Aug;12(8):822-38. doi: 10.1016/S1474-4422(13)70124-8. PMID 23867200
- [Result] Ma YJ, Fan S, Shao H, Du J, Szeverenyi NM, Young IR, Bydder GM. Use of Multiplied, Added, Subtracted and/or FiTted Inversion Recovery (MASTIR) pulse sequences. Quant Imaging Med Surg. 2020 Jun;10(6):1334-1369. doi: 10.21037/qims-20-568. PMID 32550142
- [Result] Ma YJ, Shao H, Fan S, Lu X, Du J, Young IR, Bydder GM. New options for increasing the sensitivity, specificity and scope of synergistic contrast magnetic resonance imaging (scMRI) using Multiplied, Added, Subtracted and/or FiTted (MASTIR) pulse sequences. Quant Imaging Med Surg. 2020 Oct;10(10):2030-2065. doi: 10.21037/qims-20-795. PMID 33014733
- [Result] Naganawa S, Nakane T, Kawai H, Taoka T. Lack of Contrast Enhancement in a Giant Perivascular Space of the Basal Ganglion on Delayed FLAIR Images: Implications for the Glymphatic System. Magn Reson Med Sci. 2017 Apr 10;16(2):89-90. doi: 10.2463/mrms.ci.2016-0114. Epub 2017 Jan 25. No abstract available. PMID 28123166
- [Result] Rasmussen MK, Mestre H, Nedergaard M. The glymphatic pathway in neurological disorders. Lancet Neurol. 2018 Nov;17(11):1016-1024. doi: 10.1016/S1474-4422(18)30318-1. PMID 30353860
- [Result] Hawkes CA, Hartig W, Kacza J, Schliebs R, Weller RO, Nicoll JA, Carare RO. Perivascular drainage of solutes is impaired in the ageing mouse brain and in the presence of cerebral amyloid angiopathy. Acta Neuropathol. 2011 Apr;121(4):431-43. doi: 10.1007/s00401-011-0801-7. Epub 2011 Jan 23. PMID 21259015